CLINICAL TRIAL: NCT03133260
Title: A Project to Improve the Diagnosis and Prognosis of Myocardial Injury Associated to Non Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Sandra Beltran, Anesthesiologyst deputy, MD., Parc de Salut Mar
Other Study IDs: MINSMAR
Record Dates: First submitted 2017-04-05; First posted 2017-04-28 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Myocardium; Injury
MeSH Terms: conditions — Wounds and Injuries | interventions — Aspirin; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non cardiac surgery: Determine perioperative troponin to diagnose perioperative MINS. In case of MINS acetylsalicylic acid and statins will be started if no contraindication. We will follow-up these patients for a year (including cardiologic evaluation after discharge)
  Interventions: Diagnostic Test: Troponin; Drug: Acetylsalicylic acid; Drug: Statin

INTERVENTIONS:
Diagnostic Test: Troponin — Troponin will be measured before surgery and postoperative at days 1,2 and 3.
Drug: Acetylsalicylic acid — 100mg acetylsalicylic acid will be started in case of MINS if no contraindication, it will be continued after hospital discharge. We will evaluate cardiovascular complications till 1 year after surgery
Drug: Statin — 40mg atorvastatin will be started in case of MINS if no contraindication, it will be continued after hospital discharge. We will evaluate cardiovascular complications till 1 year after surgery

SUMMARY:
Major adverse cardiovascular events are the leading cause of perioperative morbimortality in non-cardiac surgery. Perioperative myocardial infarction is usually asymptomatic, with a mortality around 10-12%.

Myocardial Injury in Noncardiac Surgery (MINS), is defined as a myocardial injury that provokes a troponin increase due to myocardial ischemia. MINS is a predictor of morbimortality at short term and at long term.

The aim of the study is to improve the diagnosis of myocardial injury after non cardiac surgery in high-risk patients, improve its treatment in case of MINS and establish prevention strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders over 45 years scheduled for non-urgent surgery with in-hospital stay of 24 hours minimum who require general and or regional anaesthesia (epidural or subarachnoidal) that have signed the inform consent who will be operated of:

  1. High-risk surgery:
* Open abdominal aortic aneurism repair
* Major vascular surgery
* Major amputations
* Carotid endarterectomy
* Duodeno-pancreatic surgery
* Hepatic resection or resection of biliary duct
* Esophagectomy
* Suprarenal resection
* Cystectomy
* Pneumonectomy

  2. Medium risk-surgery with cardiovascular risk factors (see below):
* Intraperitoneal surgery (rectum, colon, small bowel, gastric surgery)
* Peripherical angioplasty
* Endovascular aneurism repair
* Head and neck surgery
* Major orthopedic surgery (hip, knee, column)
* Major urological or gynecological surgery
* Thoracic surgery (lobectomy or atypical pulmonary resections)

  a) With 1 risk factor:
* History of coronary artery disease
* History of cerebrovascular disease (history of transient ischemic attack or stroke)
* History of congestive heart failure
* History of vascular disease

  b) With 2 risk factors:
* Diabetes mellitus with medical treatment
* Renal disease (FGE < 45 ml•min-1•1.73m2 )
* Functional capacity < 4METs
* Intraoperative blood loss >600ml

Exclusion Criteria:

* Patients without consent information
* Patients non included in the inclusion criteria

Min Age: 45 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients of both genders over 45 years scheduled for non-urgent surgery with in-hospital stay of 24 hours minimum who require general and or regional anaesthesia (epidural or subarachnoidal) for high-risk surgery or middle risk-surgery with cardiovascular risk factors.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Prevalence of myocardial injury after non cardiac surgery (MINS). | From the day of surgery until the third postoperative day
  The aim of the study is to know the prevalence of myocardial injury after non cardiac surgery in high-risk surgical patients. The investigators will perform seriated troponin on the first 3 postoperative days, if troponin value are 30ng/L or more, the investigators will evaluate if troponin increase is due to cardiac or non-cardiac etiology (patients with TEP or sepsis will be excluded). Once the non-cardiac etiology is ruled out, it will be diagnosed of MINS

SECONDARY OUTCOMES:
Percentage of MINS which corresponds to myocardial infarction | From the day of surgery until the third postoperative day
  Evaluate the percentage of MINS that corresponds to myocardial infarction. In all patients with the diagnosis of MINS the investigators will perform an ECG to evaluate ischemic changes, an echocardiogram to evaluate dyskinesias or akinesia or the presence of ischemic symptoms. If any of them are present, the investigators will diagnose the patient of acute myocardial infarction. So the investigators will compare number of patients who present a MINS with and without myocardial infarction.
Morbimortality in high-risk surgery patients until hospital discharge | From the day of surgery until hospital discharge or until 30 days after surgery in case the patient still hospitalized
  Analyze morbimortality at hospital discharge of all patients included in the study.
Compare the prognosis of patients with MINS versus patients who present a myocardial infarction versus who presented non of them. | From the day of surgery until 1 year after surgery
  To compare short and long term prognosis (hospital discharge, 30 days, 6 months and 1 year after surgery) of patients who presented MINS vs patients who presented myocardial infarction vs patients who did not presented any of them. The investigators will evaluate major cardiovascular events, non-cardiovascular complications and cardiac and all cause mortality.
Morbimortality in high-risk surgery patients 30 days after surgery | From the day of surgery until 30 days after surgery
  Analyze morbimortality at 30 days of all patients included in the study
Morbimortality in high-risk surgery patients 6 months after surgery | From the day of surgery until 6 months after surgery
  Analyze morbimortality at 6 postoperative months of all patients included in the study
Long term morbimortality in high-risk surgery patients | From the day of surgery until 1 year after surgery
  Analyze morbimortality of all patients included in the study 1 year after surgery

OTHER OUTCOMES:
Analysis and validation of risk predictors for perioperative major adverse cardiovascular events. | From the day of surgery until 1 year after surgery
  Analyse clinical risk factors for MINS, compare current MACCE clinical risk scores as predictors of MINS and develop a new score for prediction of MINS

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Beltran, MD, Principal Investigator — Anesthetist
Locations (1):
- Hospital Del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mases A, Beltran de Heredia S, Gallart L, Roman L, Bosch L, Nunez M, Rueda M, Recasens L, Sabate S. Prediction of Acute Myocardial Injury in Noncardiac Surgery in Patients at Risk for Major Adverse Cardiovascular and Cerebrovascular Events: A Multivariable Risk Model. Anesth Analg. 2023 Dec 1;137(6):1116-1126. doi: 10.1213/ANE.0000000000006469. Epub 2023 Apr 12. PMID 37043386